CLINICAL TRIAL: NCT06106217
Title: INVESTIGATION OF THE EFFECTS OF BAPNE AND QI GONG EXERCISES ON BALANCE AND QUALITY OF LIFE IN INDIVIDUALS OVER 60
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, yakup cemel, physioyherapist, Medipol University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: istanbul MUH
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Biomechanics, Anatomy, Psychology, Neuroscience, Ethnomusicology Method; qi Gong; Quality of Life; Balance
MeSH Terms: interventions — Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bapne (Experimental)
  Interventions: Other: bapne
- qi gong (Experimental)
  Interventions: Other: qi gong

INTERVENTIONS:
Other: bapne — An exercise program was created in the form of a movement sequence consisting of nine movement combinations.
  Arms: bapne
Other: qi gong — The exercise program, which was prepared in a 40-minute sequence, was arranged as 10 minutes of warm-up, 20 minutes of Qi Gong exercises, and 10 minutes of cool-down.
  Arms: qi gong

SUMMARY:
Geriatric problems develop with aging in individuals over 60 years of age. These problems include muscle weakness, balance disorders and changes in quality of life. The aim of our study is to examine the effects of BAPNE (BMe) and qi gong (QG) exercises on balance and quality of life in individuals over the age of 60. In this study, parameters such as fall risk, muscle testing, balance, functional capacity, cognitive functions, depression and sleep quality were evaluated. 56 participants were included in the study. All cases were evaluated for the first time before they were included in the study. In the initial evaluation, Itaki fall risk questionnaire, 6-minute walk test, Berg balance scale, Pittsburg sleep quality index, World Health Organization quality of life scale elderly module, Beck depression scale, mini mental state test, object flipping test, word fluency test, stroop test, muscle strength with Jtech brand myometer and balance on Libra balance board were measured. Participants were divided into groups of 2-6 people, and second assessments were made after a total of 20 sessions of BMe exercises for 6 weeks. After a 2-week rest period, the participants were included in the third assessment and included a total of 20 sessions of QG exercise over 6 weeks. At the end of 6 weeks, the fourth evaluation was made.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old or older
* Able to walk independently
* Volunteering to exercise at least 3 days a week within the scope of the research

Exclusion Criteria:

* Having an orthopedic or surgical problem that prevents walking or exercising
* Having any neurological problems
* The presence of a pulmonary, cardiac, or systemic disease that would constitute a contraindication for exercise.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Ithaki Fall Risk Questionnaire | 14 weeks
  This developed scale consists of a total of 19 risk factors, including risk factors that may cause patient falls. Risk factors were categorized as major and minor, and minor risk factors were given 1 point and major risk factors were given 5 points. Two risk levels, low and high, were determined over the total score obtained as a result of the evaluation of risk factors. In order to distinguish high-risk patients and to take necessary precautions, it is envisaged to use the "Four Leaf Clover" figure in patients at high risk of falling.
Berg Balance Scale | 14 weeks
  Berg balance scale is a valid, reliable and sensitive measurement method that measures functional balance. The test, which includes 14 functional tests and is completed in an average of 10-20 minutes, has a score between 0-4. At 0, the loss of balance is maximum, while at a value of 4, the patient is independent of balance. The maximum score of the test is 56, and the minimum score is 0. A high score indicates good functional balance.
Libra Balance Board | 14 weeks
  Balance board produced by Easytech is a computer aided balance measuring device. This device measures 42x9x42 cm and weighs 2.7 kilograms. It gives a score out of 100, 0 points the best balance and 100 points the worst balance.
Pittsburgh Sleep Quality Index | 14 weeks
  Buysse et al. It is a scale that defines good and bad sleep, developed by in 1989. A total of 24 questions, 19 of which are self-assessed, and 5 are answered by a roommate or spouse. These assess sleep duration, latency, and the frequency and severity of specific sleep-related problems. Evaluated with points between 0-3.
WHOQOL-old | 14 weeks
  It consists of 24 questions translated into Turkish as the World Health Organization quality of life module for the elderly. Validity reliability Eser S. et al. module made by; autonomy, past present and future activities, social inheritance, death-death and intimacy.

SECONDARY OUTCOMES:
Demographic information | Baseline (only in the first evaluation)
  Name, surname, date of birth, gender, address, education level of the participants who participated in the study were recorded. They were recorded in the demographic information form.
Muscle Strength Rating | 14 weeks
  Electronic myometer was used to evaluate muscle strength. Muscle strength was measured with a Jtech brand myometer. To hip flexors, extensors, abductors and adductors, knee extensors and flexors, ankle plantar and dorsi flexors, trunk extensors and abdominals, shoulder abductors, adductors, flexors and extensors, elbow flexors and extensors, wrist flexors and extensors, wrist flexor muscle and extensors will be applied. The muscle test will be performed on the dominant side for the extremities.
6 Minute Walk Test | 14 weeks
  The 6-minute walk test is one of the tests that reflects functional performance. This test is carried out in a 30-meter corridor with the dimensions of 10x40 meters. Patients are asked to walk at the highest speed they can walk for 6 minutes, but without running. The patients are encouraged verbally before and during the walk and it is ensured that they do not lose their motivation. As a result of the test, blood pressure and heart rate values, how many meters they walked in 6 minutes are recorded.
Beck Depression Scale | 14 weeks
  It is a tool used to measure the severity of depression with 21 multiple-choice questions created by Aaron T. Beck and a Turkish version of the study. The symptoms of depression show up in our emotions and our bodies. Beck depression scale measures both of these factors, thus providing a more comprehensive and accurate diagnosis.
Mini Mental Test | 14 weeks
  First, Folstein et al. The test published by Molloy and Standish in 1997 and standardized by Güngen C. et al. Turkish validity and reliability study was conducted by It is a short, useful and standardized method that can be used to determine the cognitive level globally.
Stroop Test | 14 weeks
  It consists of 60 boxes with random red, blue and green colors and 60 randomly arranged words "red", "green" and "blue" with different ink colors and different colors. The test consists of three main tasks. The time to finish the test, the number of errors and the number of spontaneous corrections are calculated. It is a complex test that evaluates multiple frontal lobe functions. In the test, the ability to perceive, the speed of processing information in the face of misleading stimuli, and the ability of the person's perception system to direct with distracting stimuli are evaluated.
Object Flip Test | 14 weeks
  It is a test in which participants try to find the coin hidden in two blue and red glasses. If the coin is known correctly 12 times in a row, the experiment is terminated. Points are given according to the number of mistakes and a maximum of 50 repetitions can be done. The lowest score in this test indicates good OFT performance.
Vocabulary Fluency Test | 14 weeks
  It is a test that takes 3 minutes in total. Participants who are asked to produce as many words as possible with the letters F, A and S are given one minute for each letter. The total number of words produced is determined as a score.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hachenberger J, Li YM, Lemola S. Physical activity, sleep and affective wellbeing on the following day: An experience sampling study. J Sleep Res. 2023 Apr;32(2):e13723. doi: 10.1111/jsr.13723. Epub 2022 Sep 18. PMID 36116773
- [Background] Zhang H, Yin L, Peng Y, Zhang G, Chen Q, Liang J, Tian S, Tong T, Liu R, Lv C, Zhao L, Liang T, Wang J, Fan L. Effect of five-elements music therapy combined with Baduanjin qigong on patients with mild COVID-19. Hong Kong J Occup Ther. 2023 Jun;36(1):31-38. doi: 10.1177/15691861231167536. Epub 2023 Apr 12. PMID 37332295
- [Background] Emek Savas DD, Yerlikaya D, G Yener G, Oktem Tanor O. Validity, Reliability and Normative Data of the Stroop Test Capa Version. Turk Psikiyatri Derg. 2020 Spring;31(1):9-21. doi: 10.5080/u23549. English, Turkish. PMID 32594475
- [Background] Figueira HA, Figueira OA, Figueira AA, Figueira JA, Polo-Ledesma RE, Lyra da Silva CR, Dantas EHM. Impact of Physical Activity on Anxiety, Depression, Stress and Quality of Life of the Older People in Brazil. Int J Environ Res Public Health. 2023 Jan 8;20(2):1127. doi: 10.3390/ijerph20021127. PMID 36673880
- [Background] Kim SG, Lim DH, Cho YH. Analysis of the reliability of the make test in young adults by using a hand-held dynamometer. J Phys Ther Sci. 2016 Aug;28(8):2238-40. doi: 10.1589/jpts.28.2238. Epub 2016 Aug 31. PMID 27630404
- [Background] Fu H, Wang L, Zhang W, Lu J, Yang M. Diagnostic test accuracy of ultrasound for sarcopenia diagnosis: A systematic review and meta-analysis. J Cachexia Sarcopenia Muscle. 2023 Feb;14(1):57-70. doi: 10.1002/jcsm.13149. Epub 2022 Dec 13. PMID 36513380
- [Background] Terrés JMP, Naranjo FJR, Martimez AC, Colomino NC. Perceptions towards wellness and life quality through body percussion BAPNE Method and cognitive stimulation in elderly people. Procedia - Social and Behavioral Sciences 152,1108 - 1113, 2014.